CLINICAL TRIAL: NCT03383653
Title: Safety Profile Following Td Vaccination in Indonesian Pregnant Woman
Status: Completed | Type: Observational
Sponsor: PT Bio Farma (Industry)
Collaborators: Indonesian Vaccine Safety Advisory Committee (Unknown)
Responsible Party: Sponsor
Other Study IDs: Td0417
Record Dates: First submitted 2017-11-01; First posted 2017-12-26 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Healthy; Pregnant
Keywords: Td Vaccine; Safety; Pregnant; Pregnant Women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess any serious systemic reaction within 30 minutes after Td immunization in pregnant woman

DETAILED DESCRIPTION:
Any local and systemic reaction after Td immunization in pregnant woman (as a routine immunization program)

ELIGIBILITY:
Inclusion Criteria:

* Healthy Pregnant Woman aged 18-39 years old
* 27-36 weeks of pregnancy
* Subject have been informed properly regarding the study and signed the informed consent form
* Subject will commit to comply with the instructions of the investigator and the schedule of the trial

Exclusion Criteria:

* Given simultaneously with other vaccines or with the interval less than 1 month with other vaccination

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant Woman
Study Population: 200 pregnant woman, 18-39 years old From provincial health primary center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Any serious adverse event occurring from inclusion until 30 minutes after the injection | 30 minutes
  local and systemic reaction

SECONDARY OUTCOMES:
Percentage of local and systemic events occurring within 72 hours after each injection | 72 hours
  any local and systemics events
Percentage of local and systemic events occurring from 72 hours up to 28 days following injection. | 72 hours - 28 days
  any local and systemics events
Percentage of serious adverse events within 28 days after injection | 28 days
  Any serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Julitasari Sundoro, MD, Principal Investigator — Indonesian Vaccine Safety Advisory Commitee
Locations (1):
- Jakarta Provincial Ministry of Health, Jakarta, Jakarta Province, Indonesia